CLINICAL TRIAL: NCT04593173
Title: Diabetic Cardiomyopathy: Diagonostic Value of 2D and 3D Left Ventricular Strains in Echocardiography in Type 2 Diabetic Patients
Brief Title: Diabetic Cardiomyopathy
Acronym: CarDiab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7905
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2020-10

CONDITIONS: Diabetic Cardiomyopathies
Keywords: Diabetes; Cardiomyopathy; Diabetic Cardiomyopathies; Type 2 diabetes; Echocardiography; Left ventricle; strain 2D and 3D
MeSH Terms: conditions — Diabetic Cardiomyopathies; Diabetes Mellitus; Cardiomyopathies; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetes represents one of the 10 leading causes of death in the world and concerns 5% of the French population (> 3.3 million patients). About 30% of diabetic patients will develop heart failure. The specific and early identification of diabetic cardiomyopathy at a subclinical stage (asymptomatic patients with normal LVEF) will thus make it possible to predict the risk of the onset of heart failure and to strengthen their monitoring and further adapt their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Type 2 diabetic and hypertensive subjects, cardiac asymptomatic, without myocardial ischemia documented by Dobutamine stress ultrasound (ESD), having at least 1 additional CV risk factor among: dyslipidemia, active or stopped smoking for less than 3 years, family history (1st degree relationship) of major CV accident before age 60, obliterating arteriopathy of the lower limbs and / or carotid atheroma, or proteinuria.
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion Criteria:

* Patient who expressed his opposition to participating in the study
* Valvular heart disease (moderate to severe valve disease), hypertrophic or dilated (MVGi> 95 g / m2 in women and MVGi> 115 g / m2 in men), chronic pulmonary;
* History of cardiotoxic chemotherapy;
* Subject under legal protection, under guardianship or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic and hypertensive patients, treated in the Internal Medicine and Diabetology Services of Strasbourg University Hospitals, between 04/15/2015 to 04/30/2019.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of Value of 2D and 3D Left Ventricular Strains in Echocardiography in Type 2 of diabetic Patients | The files analysed retrospectily from April 15, 2015 to April 30, 2019 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Physiologie et d'Explorations Fonctionnelles, Strasbourg, Starsbourg, France